CLINICAL TRIAL: NCT00083408
Title: UARK 99-016, A Phase II Trial of Combination Bisphosphonate and Anti-Angiogenesis Therapy With Pamidronate and Thalidomide in Patients With Multiple Myeloma and Poor Hematopoietic Stem Cell Reserve
Brief Title: Combination Bisphosphonate and Anti-Angiogenesis Therapy With Pamidronate and Thalidomide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UARK 99-016
Record Dates: First submitted 2004-05-24; First posted 2004-05-25 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Pamidronate; Thalidomide; refractory myeloma; bisphosphonates; Aredia
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Pamidronate; Thalidomide

INTERVENTIONS:
Drug: Pamidronate
Drug: Thalidomide

SUMMARY:
The purpose of this research is to study how helpful the combination of thalidomide and Pamidronate is in controlling multiple myeloma and to study any side effects that may be experienced.

DETAILED DESCRIPTION:
Recently, laboratory research found that thalidomide can inhibit the formation of new blood vessels that are necessary for the growth and spread of cancer. In order to grow and increase in size, tumors require new blood vessels to supply them with the necessary blood to grow. If we can prevent these new blood vessels feeding the tumor from being formed by using thalidomide we might slow or stop the growth of the tumor. This concept is called "anti-angiogenesis". It is hoped that thalidomide will slow or stop the growth myeloma. However, it cannot be guaranteed that you will benefit if you take part in this study. The treatment you receive may even be harmful.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of Multiple myeloma with poor hematopoietic reserve (platelet count <100,000 OR inability to collect adequate PBSC to support autologous transplant (4X106 CD34+cells/kg OR WBC <2,000)
* Patients must not be eligible for UARK 98-035
* Patients must be at least 6 weeks beyond previous chemotherapy
* All patients must be informed of the investigational nature of this study and must sign a written informed consent in accordance with UAMS Human Research Advisory Committee and federal guidelines

Exclusion Criteria:

* Prior bisphosphonate therapy within 30 days prior to study entry
* Serum creatinine > 5 mg/dl, ascites, or serum direct bilirubin > 2.5 mg/dl
* Prior plicamycin or calcitonin within 2 weeks of study entry
* Severe cardiac disease, unstable thyroid disease, or epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 1998-03; Study Completion 2005-05

PRIMARY OUTCOMES:
To evaluate the effectiveness of combination treatment with Thalidomide and Pamidronate in patients with refractory myeloma and poor hematopoietic stem cell reserve. Effectiveness will be based on the estimate of the objective response rate (CR + PR).

SECONDARY OUTCOMES:
To compare the effect of these agents on disease parameters, specifically on time to disease progression and overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Fassas, M.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- See also: Myeloma Institute for Research & Therapy website — http://myeloma.uams.edu